CLINICAL TRIAL: NCT00524004
Title: Protective Efficacy of Orally Delivered Bovine Immunoglobulin, Specific for CS17 Fimbriae and CS17 Minor Fimbrial Adhesin CsbD Against Challenge With a CS17 Strain of Enterotoxigenic Escherichia Coli (ETEC)
Brief Title: Safety and Efficacy of Bovine Milk Immunoglobulin Against CS17 and CsbD
Acronym: BIgGII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Naval Medical Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, August Louis Bourgeois, Senior Scientist, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 233; WIRB Approval Number 20062031 (Other: WIRB); W81XWH-04-1-0067 (Other Grant/Funding Number: Department of the Army)
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Travelers' Diarrhea
Keywords: Passive immunization, Bovine Milk Immunoglobulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Anti-CsbD Bovine IgG (Experimental): Anti CsbD Bovine Milk Immunoglobulin
  Interventions: Other: Placebo; Biological: Anti-CS17 Bovin IgG
- Placebo (Experimental): Lacto-free milk supplement
  Interventions: Biological: Anti-CS17 Bovin IgG
- Anti-CS17 Bovin IgG (Experimental): Anti-CS17 Bovin Milk Immunoglobulin
  Interventions: Biological: Anti-CsbD Bovine IgG; Biological: Anti-CS17 Bovin IgG

INTERVENTIONS:
Biological: Anti-CsbD Bovine IgG — Three times a day for seven days
  Other Names: Experimental
  Arms: Anti-CS17 Bovin IgG
Other: Placebo — Three times a day for seven days
  Other Names: Lacto-Free milk supplement
  Arms: Anti-CsbD Bovine IgG
Biological: Anti-CS17 Bovin IgG — Three times a day for seven days
  Other Names: Experimental

SUMMARY:
This is a Phase II, randomized, double-blind, placebo-controlled study designed to investigate whether hyperimmune bovine milk IgG products specific for CsbD and CS17, protect subjects against diarrhea upon challenge with a CS-17-ETEC strain LSN03-016011/A. The study will also evaluate safety and tolerability of these bovine milk IgG products and describe the immune responses following challenge.

The primary study objectives are: 1) Assess safety of the anti-CsbD and anti-CS17 bovine milk IgG among healthy adult volunteers when orally administered three times a day over 7 days. 2) Determine efficacy of the anti-CsbD bovine milk IgG preparation against ETEC diarrhea upon challenge with CS17-ETEC, and 3)Determine efficacy of the anti-CS17 bovine milk IgG preparation against ETEC diarrhea upon challenge with CS17-ETEC. A secondary objective is to determine efficacy of the anti-CsbD and anti-CS17 bovine milk IgG preparations against moderate to severe ETEC diarrhea upon challenge with CS17-ETEC.

DETAILED DESCRIPTION:
The primary study objectives are: 1) Assess safety of the anti-CsbD and anti-CS17 bovine milk IgG among healthy adult volunteers when orally administered three times a day over 7 days. 2) Determine efficacy of the anti-CsbD bovine milk IgG preparation against ETEC diarrhea upon challenge with CS17-ETEC, and 3)Determine efficacy of the anti-CS17 bovine milk IgG preparation against ETEC diarrhea upon challenge with CS17-ETEC. A secondary objective is to determine efficacy of the anti-CsbD and anti-CS17 bovine milk IgG preparations against moderate to severe ETEC diarrhea upon challenge with CS17-ETEC.

STUDY DESIGN This is a Phase II, randomized, double-blind, placebo-controlled study designed to investigate whether hyperimmune bovine milk IgG products specific for CsbD and CS17, protect subjects against diarrhea upon challenge with a CS-17-ETEC strain LSN03-016011/A. The study will also evaluate safety and tolerability of these bovine milk IgG products and describe the immune responses following challenge.

Subjects (N=39) will be randomized into three groups receiving anti-CS17 bovine milk IgG, anti-CsbD bovine milk IgG, or a placebo control (a commercially available lactose-free infant formula called LactoFree® Lipil®) on study day -2. Subjects will receive three doses a day of the test article 15 minutes (range 10 - 25 minutes) after each of their three daily meals (breakfast, lunch and dinner) for a period of 7 days (i.e., from study day -2 to study day 4). The study will be divided into two cohorts, An initial cohort of 9 subjects (3 per treatment group), will be admitted to the General Clinical Research Center (GCRC) of the Johns Hopkins Hospital for the initial testing of the bovine milk IgG products. A second cohort of 30 subjects will then be admitted to the Bayview inpatient facility to complete the prophylaxis study. Logistical considerations and/or withdrawals or disqualifications prior to admission or after randomization, but prior to receiving the ETEC challenge, may require a third cohort to be admitted to either of these facilities. Allowing for these contingencies, the minimum number of subjects to be challenged with ETEC is 33 total and the maximum number of subjects will be 42. The GCRC Project Review Committee will review the protocol prior to subject admission at the GCRC. A brief description of the two inpatient facilities to be used in this study is provided in Section 6.1.2. Unit doses of the test article powders (as detailed in Table 5) will be suspended in 150 mL of water containing 2 grams of sodium bicarbonate buffer. Doses of the test articles/placebo will be prepared by study staff under the supervision of the research pharmacist. The study staff involved in dose preparation will not be collecting clinical data on subjects. On the fourth day of the inpatient phase (study day 0), after their morning meal and receipt of test article/placebo, subjects will be given 120mL of sodium bicarbonate buffer to neutralize their stomach acidity. About 1 minute later they will ingest a dose of CS17-ETEC strain LSN03-016011/A (5 X 109 cfu) diluted in 30 ml sodium bicarbonate buffer. Subjects will continue to receive three doses a day of the test articles/placebo until study day 4. Subjects meeting preset criteria will be treated with antibiotics within 24 hours of determination by the investigator and test article/placebo administration will be discontinued with initiation of treatment. Subjects who do not receive early antibiotic treatment will start antibiotic treatment on study day 5. Routine discharge is scheduled for day 7, when most subjects are expected to meet the discharge criteria of: they feel well(clinical symptoms resolved or resolving and have taken at least one dose of antibiotic and have 1 stool culture negative for the challenge strain. Subjects may be discharged earlier than day 7 on a case-by-case basis if they meet discharge criteria. The duration of the active study period is approximately seven months, encompassing up to 6 and 1/2 weeks of screening/enrollment, 4 weeks of the inpatient/outpatient phase when data and samples will be collected, 12 weeks for immunology assays, and 2 months for analysis and report.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 45 years of age
2. General good health, without significant medical illness, abnormal physical exam findings or clinically significant lab abnormalities, as determined by the PI
3. Demonstrate comprehension of the protocol procedures and knowledge of ETEC illness by passing a written exam (pass grade ≥ 70%)
4. Willing to participate after informed consent obtained
5. Available for all planned follow-up visits
6. Negative serum pregnancy test at screening; on the day of admission to the inpatient phase for female subjects of childbearing potential. Females of childbearing potential must agree to use an efficacious hormonal or barrier method of birth control during the study. Abstinence is acceptable. Female unable to bear children must have this documented (e.g., tubal ligation or hysterectomy).

Exclusion Criteria:

1. Presence of significant medical conditions such as psychiatric conditions, gastrointestinal disease (such as peptic ulcer, active gastritis or gastroesophageal reflux disease, inflammatory bowel disease), alcohol or illicit drug abuse/dependency, or lab abnormalities which in the opinion of the investigator precludes participation in the study
2. Immunosuppressive illness or IgA deficiency (below the normal limits)
3. Positive serology results for HIV or HCV antibodies, or HBsAg
4. Significant abnormalities in screening hematology, serum chemistry, urinalysis or EKG (EKG in subjects ≥ 40 years), as determined by the PI
5. Allergy to fluoroquinolones, trimethoprim-sulfamethoxazole, or ampicillin/penicillin (excluded if allergic to 2 of 3)
6. Fewer than 3 stools per week or more than 3 stools per day on a regular basis.
7. History of diarrhea in the 2 weeks prior to planned inpatient phase
8. Regular use of laxatives, antacids, or other agents to lower stomach acidity (regular = at least weekly)
9. Use of antibiotics during the 7 days before dosing or proton pump inhibitors, H2 blockers, or antacids within 48 hours of dosing (bovine milk IgG).
10. Travel to countries where ETEC or cholera infection is endemic (most of the developing world) within 2 years prior to bovine milk IgG dosing
11. History of vaccination for or ingestion of ETEC, cholera, or LT toxin.
12. Stool culture (collected no more than 1 week prior to admission) positive for ETEC or other bacterial enteric pathogens (including Salmonella, Shigella and Campylobacter)
13. Use of any investigational drug or any investigational vaccine within 30 days preceding the first dose of test article/placebo, or planned use during the active study period
14. Clinical history of lactose intolerance or allergy to milk or milk products
15. Use of any medication known to affect the immune function (e.g., corticosteroids) within 30 days preceding the first dose of test article/placebo, or planned use during the active study period. (Topical and intra-articular steroids will not exclude subjects.)
16. Inability to tolerate an over-the-counter, lactose-free, infant, powder formula suspended in 150 mL sodium bicarbonate buffer (based on requirement for frequent dosing) Subjects will receive a dose of the test article 3 times daily 15 minutes (range 10-25 minutes) after each meal for 7 days. The dose will consist of 2.4 gm anti-CS17 bovine milk IgG, 2.3 gm anti-CsbD bovine milk IgG or 2.8 gm LactoFree® powder suspended in 150 mL of water containing 2 grams of sodium bicarbonate buffer.

    * Breakfast and 1st daily dose of test article as described above
    * Following a 90-minute fast, subjects will ingest 120 ml of sodium bicarbonate buffer to neutralize stomach acidity.
    * One minute later (up to 2 minutes) subjects will ingest the CS17-ETEC challenge inoculum diluted in 30ml sodium bicarbonate buffer.
    * Fifteen minutes (range: 10-25 minutes) after drinking the CS17-ETEC inoculum, subjects will ingest the second (Day 0) dose of bovine milk IgG test article or placebo.
    * No IgG test articles will be administered immediately following lunch on the day of challenge.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-01-30 (Actual); Primary Completion 2007-10-26 (Actual); Study Completion 2007-10-26 (Actual)

PRIMARY OUTCOMES:
Prevention of ETEC diarrhea | 120 hours after challenge

SECONDARY OUTCOMES:
Prevention of moderate to severe ETEC diarrhea | 120 hours after challenge

CONTACTS AND LOCATIONS:
Overall Officials: Robin McKenzie, M.D., Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- United States (2):
  - Center for Immunization Research, Baltimore, Maryland
  - Johns Hopkins Bayview Medicial Center, Inpatient Unit, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Savarino SJ, McKenzie R, Tribble DR, Porter CK, O'Dowd A, Sincock SA, Poole ST, DeNearing B, Woods CM, Kim H, Grahek SL, Brinkley C, Crabb JH, Bourgeois AL. Hyperimmune Bovine Colostral Anti-CS17 Antibodies Protect Against Enterotoxigenic Escherichia coli Diarrhea in a Randomized, Doubled-Blind, Placebo-Controlled Human Infection Model. J Infect Dis. 2019 Jul 2;220(3):505-513. doi: 10.1093/infdis/jiz135. PMID 30897198